CLINICAL TRIAL: NCT00050921
Title: Improving Immune Reconstitution With Growth Hormone in HIV-infected Subjects With Incomplete CD4+ Lymphocyte Restoration on Highly Active Antiretroviral Therapy (HAART)
Brief Title: Administration of Growth Hormone to Increase CD4+ Count in Patients Taking Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5174; ACTG A5198s; 10092 (Registry Identifier: DAIDS ES Registry Number); ACTG A5174
Record Dates: First submitted 2002-12-30; First posted 2003-01-01 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Infections; CD4 Lymphocyte Count; Antiretroviral Therapy, Highly Active; Growth Hormone; Cell Division; CD4-Positive T-Lymphocytes; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Human Growth Hormone; Hepatitis A Vaccines; keyhole-limpet hemocyanin

INTERVENTIONS:
Drug: somatropin
Biological: Hepatitis A virus, inactivated
Drug: Keyhole-Limpet Hemocyanin

SUMMARY:
This study is designed to evaluate the ability of growth hormone (GH, also known as somatropin) to increase CD4+ cell counts in patients taking anti-HIV drugs. The study is targeted toward patients with low levels of HIV who continue to have low CD4+ cell counts.

DETAILED DESCRIPTION:
After initiation of HAART, many HIV infected patients have significant improvement in CD4+ levels. However, some patients continue to have low CD4+ counts (< 350 cells/mm3) despite adequate viral suppression. The purpose of this study is to determine whether administration of GH will increase naïve CD4+ production. Further, the study will assess whether an increase in naïve CD4+ production will lead to increases in antigen-specific CD4+ and CD8+ T cells.

Patients enrolled in this study will be randomized to one of two groups. Patients in both groups will continue their present HAART regimen for the duration of the study. Group A patients will receive daily subcutaneous injections of GH for 48 weeks. Group B participants will receive no additional therapy for 24 weeks, and will then receive daily subcutaneous GH injections during Weeks 24-28 of the study. Both groups will receive immunocyanin (keyhole-limpet hemocyanin) injections at Weeks 16 and 20 and hepatitis A vaccination at Weeks 40 and 44. At the conclusion of Week 48, all patients will discontinue GH therapy while maintaining their HAART regimen. Patients will then be followed for an additional 24 weeks.

Patients may be asked to participate in a substudy to measure the size of the thymus in people taking GH. Patients in the substudy will have a noncontrast CT scan of the chest before beginning GH therapy and again after 24 weeks of GH therapy.

ELIGIBILITY:
Inclusion Criteria

* HIV positive
* Minimum of 1 year of treatment with HAART
* CD4+ cell count <350 cells/mm3
* HIV-1 RNA <400 copies/ml for 6 months prior to study entry
* Acceptable methods of contraception

Exclusion Criteria

* Serious medical illness requiring hospitalization within 14 days prior to study entry
* Pregnant or breast-feeding
* Taking certain medications
* Allergy to r-hGH, hepatitis A vaccine, KLH, or their formulations, including allergies to shellfish
* Active drug or alcohol dependence
* Diabetes or uncontrolled hyperglycemia
* Uncontrolled hypertension
* History of carpal tunnel syndrome
* Active neoplasm requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Smith, M.D., MPH, Study Chair — Rush Medical College of Rush University
Locations (13):
- United States (13):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Univ. of Texas Southwestern Med. Ctr., Amelia Court Continuity Clinic, Dallas, Texas

REFERENCES:
- [Background] Connick E, Lederman MM, Kotzin BL, Spritzler J, Kuritzkes DR, St Clair M, Sevin AD, Fox L, Chiozzi MH, Leonard JM, Rousseau F, D'Arc Roe J, Martinez A, Kessler H, Landay A. Immune reconstitution in the first year of potent antiretroviral therapy and its relationship to virologic response. J Infect Dis. 2000 Jan;181(1):358-63. doi: 10.1086/315171. PMID 10608789
- [Background] Smith KY, Valdez H, Landay A, Spritzler J, Kessler HA, Connick E, Kuritzkes D, Gross B, Francis I, McCune JM, Lederman MM. Thymic size and lymphocyte restoration in patients with human immunodeficiency virus infection after 48 weeks of zidovudine, lamivudine, and ritonavir therapy. J Infect Dis. 2000 Jan;181(1):141-7. doi: 10.1086/315169. PMID 10608760
- [Background] Vigano A, Vella S, Saresella M, Vanzulli A, Bricalli D, Di Fabio S, Ferrante P, Andreotti M, Pirillo M, Dally LG, Clerici M, Principi N. Early immune reconstitution after potent antiretroviral therapy in HIV-infected children correlates with the increase in thymus volume. AIDS. 2000 Feb 18;14(3):251-61. doi: 10.1097/00002030-200002180-00007. PMID 10716501
- [Background] Schambelan M, Mulligan K, Grunfeld C, Daar ES, LaMarca A, Kotler DP, Wang J, Bozzette SA, Breitmeyer JB. Recombinant human growth hormone in patients with HIV-associated wasting. A randomized, placebo-controlled trial. Serostim Study Group. Ann Intern Med. 1996 Dec 1;125(11):873-82. doi: 10.7326/0003-4819-125-11-199612010-00002. PMID 8967667
- [Background] Napolitano LA, Lo JC, Gotway MB, Mulligan K, Barbour JD, Schmidt D, Grant RM, Halvorsen RA, Schambelan M, McCune JM. Increased thymic mass and circulating naive CD4 T cells in HIV-1-infected adults treated with growth hormone. AIDS. 2002 May 24;16(8):1103-11. doi: 10.1097/00002030-200205240-00003. PMID 12004268